CLINICAL TRIAL: NCT06232395
Title: Early Detection and Post-operative Monitoring of Gastric Cancer Using Circulating DNA in Blood Samples
Brief Title: Early Detection and Post-operative Monitoring of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Suzhou Huhu Health & Technology Inc. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2311285-6
Record Dates: First submitted 2024-01-17; First posted 2024-01-30 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Human Papillomavirus DNA Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected from each study participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- malignant group: Subjects diagnosed with gastric cancer.
  Interventions: Diagnostic Test: DNA test
- non-malignant group: Healthy individuals and subjects with gastritis, gastric ulcer, gastric polyp or other benign gastric diseases.
  Interventions: Diagnostic Test: DNA test

INTERVENTIONS:
Diagnostic Test: DNA test — circulating DNA test

SUMMARY:
This study is to determine the performance of non-invasive new multi-target biomarkers in the early detection and post-operative monitoring of gastric cancer.

DETAILED DESCRIPTION:
This study aims to develop and validate a new non-invasive detection method for early detection and postoperative monitoring of gastric cancer in the blood. Sensitivity, specificity, accuracy, ROC curve area, positive predictive value, and negative predictive value of the new biomarkers in the diagnosis of gastric cancer will be compared with that of tumor biomarkers CA19-9, CEA, and CA72-4. Blood will also be collected at various time points post-operatively. The investigators will determine whether these new biomarkers can be used as prognostic biomarkers to predict tumor recurrence and metastasis. The investigators will also determine whether these new biomarkers detect tumor recurrence and metastasis earlier than methods currently used in the clinic such as imaging and tumor biomarkers CA19-9, CEA, and CA72-4.

This study is a prospective and multi-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age over 18.
2. Subject has stomach discomfort, and seek medical attention at the Gastric Surgery Department of our center.
3. Subject has or will have gastroscopy and/or pathological examination results at this center.
4. Subject must be able to fully understand the informed consent form and be able to personally sign it.

Exclusion Criteria:

1. Subject has serious heart, liver, kidney dysfunction, or mental illness.
2. Subject diagnosed previously with any kind of malignant tumor.
3. Subject is known to be infected with HIV or other related diseases (considering interference from the use of immune drugs).
4. Subject is receiving targeted drugs, immunosuppressants, immunomodulators, and biological therapies.
5. Researchers believe that subject is not suitable for enrollment.
6. Subject can not supply sufficient sample to complete this experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects age over 18, regardless of gender or region, and those who meet the inclusion criteria for this clinical trial, are eligible to enroll at the designated clinical sites. More than 1197subjects are targeted to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 1197 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
The performance of the new detection system for gastric cancer (GC) detection | 2 years
  Evaluate sensitivity, specificity, accuracy, ROC curve area, positive predictive value, and negative predictive value of the new biomarker for the diagnosis of gastric cancer.
The performance of the new biomarkers in the post-operative monitoring of gastric cancer | 2 years
  Determine whether the new detection system can detect tumor recurrence and metastasis earlier than imaging and tumor marker CA19-9, CEA, and CA72-4.

SECONDARY OUTCOMES:
Compare the performance of the new biomarkers for GC detection with the conventional tumor markers | 2 years
  Determine whether the performance of the new biomarker detection system is better than that of tumor markers CA19-9, CEA, and CA72-4 in the diagnosis of gastric cancer.
The performance of the new biomarkers as prognostic biomarkers | 2 years
  Determine whether the new biomarkers cancer serve as prognostic biomarkers to predict tumor recurrence and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No